CLINICAL TRIAL: NCT06461741
Title: Integrated Dual-task EMG Biofeedback Balance Training to Improve Balance in Individuals Living with Multiple Sclerosis
Brief Title: EMG Biofeedback Training to Improve Balance in Individuals with Multiple Sclerosis
Acronym: MSBAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS Balance Study
Record Dates: First submitted 2024-06-10; First posted 2024-06-17 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
Keywords: Balance; Falls
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Dual-task EMG Biofeedback Training (EMG-BF) (Experimental): Participants will engage in EMG-BF for 30 minutes 3 times per week for 6 weeks for a total of 18 sessions. Our novel EMG Biofeedback training system can be adapted to a training objective by planning 3 to 5 movements and placing sensors over muscles that must be active when the user adheres to the correct movement form. For our training we use right or left torso shift with knee bend, and right or left hand opening, and place sensors over left and right vastus lateralis and left and right extensor digitorum superficialis muscles.
  Each movement corresponds to a specific videogame command. To introduce cognitive challenge, we randomly shuffle the game command assigned to each movement at the beginning of every session. This will require the user to choose the appropriate movement to trigger the intended game input while suppressing incorrect movements. We use the puzzle game, Tetris, which requires spatial reasoning and planning under increasingly tight time constraints.
  Interventions: Device: Integrated Dual-task EMG Biofeedback Training (EMG-BF)
- Traditional Balance Exercise Training (BAL-EX) (Active Comparator): Participants will perform 7 balance exercises traditionally prescribed by physiotherapists. The first is a heel/toe square exercise where the trainee lifts their right toe and left heel, then their left toe and right heel, then both heels, then both toes. The 2nd exercise involves maintaining tandem stance while static, then moving the arms, then looking up and down, then looking left and right. The 3rd exercise is lateral stepping where the individual steps with one foot out to the side and then bring the foot back to the starting stance. The 4th exercise is a golfer's lift where the person slowly leans forward while extending one leg straight behind and touches the seat of a chair placed opposite. The 5th exercise is extended-duration single leg stands and exercises 6 and 7 are back and side leg raises, respectively. The exercise sequence will repeat until 30 minutes has expired. Sessions are repeated 3 times per week for 6 weeks, for 18 sessions.
  Interventions: Behavioral: Traditional Balance Exercise Training (BAL-EX)

INTERVENTIONS:
Device: Integrated Dual-task EMG Biofeedback Training (EMG-BF) — The intervention is an exercise training that is facilitated by feedback derived from electrical muscle activity measured through electromyography (EMG). An EMG Biofeedback software uses a machine learning algorithm to identify the desired movements and reinforce them by displaying feedback on a computer monitor in the form of videogame control. The EMG acquisition hardware must have at least 4 sensor channels and a sampling rate of >1KHz. Other than these specifications, any generic EMG amplifier can be used. The effect of the "device" is therefore primarily defined by the software. An in-depth description of the software and hardware systems is published in the cites study, "An EMG-Based Biofeedback System for Tailored Interventions Involving Distributed Muscles". In this trail is the Explore+ ExG amplifier which is sold by Mentalab.
  Arms: Integrated Dual-task EMG Biofeedback Training (EMG-BF)
Behavioral: Traditional Balance Exercise Training (BAL-EX) — This intervention is a time-matched active comparator for the EMG-BF intervention. A sequence of seven traditional, balance exercises, taking 1-3 minutes each, is repeated for a total of 30 minutes on each of 18 sessions in the 6-week intervention period. The exercises are ones that challenge the coordination and strength of postural muscles in the presence of various vestibular stimuli. The specific exercises are described in the Arm description.
  Arms: Traditional Balance Exercise Training (BAL-EX)

SUMMARY:
The goal of this clinical trial is to test the impact of a novel dual-task EMG Biofeedback training method for improving balance in individuals living with multiple sclerosis. The main question[s] it aims to answer are:

* Does dual-task EMG biofeedback training deliver lasting balance benefits up to 3 months following the intervention?
* Are the benefits greater than those for participation in traditional balance training exercises?
* Do the benefits vary with the severity of disability?

Participants will receive either EMG Biofeedback (EMG-BF) training or traditional balance exercise (BAL-EX) training. Both treatments involve three 30-minute sessions of the training every week for 6 weeks (18 sessions). During the sessions, participants in the EMG-BF treatment group will perform targeted exercises using feedback from adhesive (sticker) sensors on their arms and legs. Participants in the BAL-EX treatment group will following an instructor through balance training movements that are traditionally prescribed by physiotherapists to improve balance. Measurements will be taken at the beginning of the study, after six weeks of training, and three months after the end of training.

Researchers will compare the groups to see if balance and related outcomes are improved more by 6-weeks of EMG-BF training than BAL-EX.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years with a formal diagnosis of MS.
* Participants must be ambulatory and report problems with walking and/or balance.
* Have stable disease with no relapses in the last 3 months.
* Agreement to not introduce or change the dosage of pharmaceutical treatments during the study period. This includes intramuscular injections (e.g., Botox), intravenous, and orally administered drugs.
* Agreement to maintain the frequency, duration and intensity of physical therapy or any alternate therapies (e.g., massage, osteopathic, chiropractic, etc.) for the duration of the trial.

Exclusion Criteria:

* Unable to follow instructions due to cognitive deficit or language barrier
* Presence of visual disorders that prevent meaningful interaction with the intervention interface.
* Unable to maintain stable pharmaceutical treatment for the duration of the study.
* Unable to maintain the frequency, duration and intensity of physical therapy or alternate therapies outside of the trial for the duration of the trial.
* Received Botox treatment within 3 months of the onset of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Mini-Balance Evaluation Systems Test (Mini-BESTest) | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  A sensitive, reliable, and valid 14-item scale that assesses dynamic balance. It includes components evaluating anticipatory postural adjustments, responses to perturbation, sensory orientation, and dynamic stability during gait. The total score ranges from 0 ("no balance") to 28 ("complete balance").

SECONDARY OUTCOMES:
Limits of Stability (LoS) | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  Assesses the ability of an individual to control the center of pressure (COP) on a force platform within their base of support. Subjects are instructed to move a cursor indicating their COP away from the center of their base of support in all directions using feedback provided on a computer monitor. The feedback includes a representation of the force plate and the COP which paints the area covered by its movements. The goal communicated to the subject is to create the largest coverage area possible without lifting their feet off the plate. Total and quadrant-specific areas (i.e., Total, Front Left, Front Right, Back left, and Back Right) are measured in cm2. These measures are reliable, and published reference values exist.
Sway in Quiet Stance (QS) | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  Assesses the movement of the participants center of center of pressure (COP) while standing on a force platform with hands on hips. The mean length in cm of the path traveled by the COP during the last 3 of 4 total subsequent 20s trials (one practice trial) is the outcome of interest. The test is repeated with eyes open, and eyes closed. This assessment is valid and reliable.
Timed 25ft Walk Test (T25WT) | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  Participants start at a line on the floor and are instructed to "walk as quickly as possible but safely" beyond the second line 25 feet away. The time is recorded in seconds beginning with the first heel strike beyond the start line and ending with the first heel strike after the second line, two trials are performed with the faster time used for the analysis. This assessment is valid and reliable.
Activities-specific Balance Confidence (ABC) scale | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  A patient-reported questionnaire regarding balance confidence during 16 everyday activities. The ABC scale is quick and easy to administer and has demonstrated good reliability, validity, and sensitivity in MS populations.
12-item Subjective Walking Scale (SWS-12) | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  A 12-item questionnaire regarding the effect of the respondent's "condition" on their walking in the last two weeks. The questions are adapted from the MS walking scale, which is a valid and reliable measurement tool.
Short-Form 36 Health Survey (SF-36) | It will be measured at baseline, 6 weeks of training, and 3 months after the end of training (18 weeks from baseline)
  A popular health-related quality of life measure with 36 items, 8 scales, and physical and mental summary measures. The scales are physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), role-emotional (RE), social functioning (SF) and mental health (MH). The summary scores are the physical health composite summary (PCS) and the mental health composite summary (MCS). The SF-36 is valid and reliable.
Fall and Near-Fall Frequency | Participant will keep the fall diary from 2 weeks before the first training session to the end of the study, 20 weeks later.
  Fall diaries are a simple and effective means to measure falls. Each participant with record falls and near-falls in a calendar by marking "F" or "NF" on the day of a fall. For each fall, participants fill a short form providing information about the cause, any injuries, or hospitalization as the result of the fall.

OTHER OUTCOMES:
Visual Analog Scales (VAS) | The weekly 3-session average will be assessed for week 1, 2, 3, 4, 5 and 6. the average across all six weeks (18 sessions) will be assessed.
  At the end of every session participants make a vertical mark on a 10-centimeter horizontal line representing a continuum between "Strongly Disagree" (0 cm) and "Strongly Agree" (10 cm). The midpoint of the line (5 cm) represents "Neither Agree nor Disagree". VAS measurements are accurate and precise. Participants will respond to VAS scales with the following prompts:
  * I enjoyed the training.
  * The training was challenging.
  * I put forth a great deal of effort.
  The average of VAS values provided in each week (3 sessions per week) of participation, and across the entire 6 weeks of training (18 sessions) will be assessed.
Enjoyment Scale (ES) | 6 weeks of training.
  Participants will respond to 5 statements adapted from a usability questionnaire developed by Ona and colleagues. For each question, responses are provided on a 10-point scale whereby 1 represents 'strongly disagree' and 10 is 'strongly agree'. The response to each statement is summed for a total of out 50.
  Statements will include:
  1. The training meets a real need.
  2. The training is intuitive and easy to understand.
  3. I will continue to use the access the training in the future if it is available.
  4. The difficulty of the training was adequate.
  5. The training sessions were enjoyable.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toepp SL, Mohrenschildt MV, and Nelson AJ. An EMG-Based Biofeedback System for Tailored Interventions Involving Distributed Muscles. IEEE Sensors Journal. 2024; 23(22): 28095-28109.
- See also: Link to the above cited work, which describes the EMG Biofeedback approach used in this trial. — https://ieeexplore.ieee.org/abstract/document/10287258?casa_token=C8XT6K3ISBcAAAAA:igNnzXFEROBb6locxsy5kjieEJx9GKsnXQ3e6oXcuhwitj-61wUvy4en5SKDKwrU41UlmUr0cg